CLINICAL TRIAL: NCT06144684
Title: A Two-Part First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Subcutaneous Doses of GUB014295 in Lean to Overweight or Obese But Otherwise Healthy Men and Women
Brief Title: A Two-Part First-In-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GUB014295
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GUC17-01; 1008236 (Other: MHRA (IRAS))
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Overweight
Keywords: Weight management
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: This phase 1 study, will be conducted to assess the safety, tolerability, and pharmacokinetics (PK) of single and multiple ascending subcutaneous doses of GUB014295
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study; each cohort will include matching placebo and active drug solutions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo solution
  Interventions: Drug: GUB014295-PLACEBO
- GUB014295 (Active Comparator): GUB014295 solution 5 mg/mL
  Interventions: Drug: GUB014295

INTERVENTIONS:
Drug: GUB014295 — GUB014295 is a long-acting amylin analogue in development, a single subcutaneous dose is administered in part 1, multiple doses administered in part 2 of the study
  Other Names: GUBamy
  Arms: GUB014295
Drug: GUB014295-PLACEBO — GUB014295-PLACEBO is matching GUB014295 in appearance, a single subcutaneous dose is administered in part 1, multiple doses administered in part 2 of the study
  Arms: Placebo

SUMMARY:
This is a two-part, single centre, double-blind (within cohorts), randomised, placebo-controlled, single (Part 1) and multiple (Part 2) ascending subcutaneous dose study in lean to overweight or obese but otherwise healthy men (Part 1) and men and non-pregnant, non-lactating women (Part 2). The primary objective is to assess the safety and tolerability. Secondary objectives are to characterize the pharmacokinetics (PK) and to investigate pharmacodynamic effects.

DETAILED DESCRIPTION:
This is a phase 1 clinical trial of a new long-acting amylin analogue GUB014295 in two parts.

Trial design: Part 1 is a double-blind (within cohorts), randomised, placebo-controlled, single ascending dose (SAD) study. It is planned to enrol 4 cohorts of 8 subjects (Regimens A, B, C and D), with 2 additional optional cohorts of 8 subjects (Regimens E and F). Part 2A is a double-blind (within cohorts), randomised, placebo-controlled, multiple ascending dose (MAD) study. It is planned to enrol 2 cohorts of 8 subjects (Regimens G and H). Part 2B is a double-blind (within cohorts), randomised, placebo-controlled, MAD study.

It is planned to enrol 3 cohorts of 12 subjects (Regimens I, J and K). Part 2C is a double-blind (within cohorts), randomised, placebo-controlled, MAD study. It is planned to enrol 2 cohorts of up to 12 subjects (Regimens L and M).

The primary objective is to assess the safety and tolerability of a new long-acting amylin-analogue GUB014295. Secondary objectives are to characterize the pharmacokinetics (PK) of the long-acting amylin-analogue GUB014295 and to investigate if the long-acting amylin-analogue GUB014295 has possible pharmacodynamic effects measured as weight changes and changes in gastric emptying (paracetamol concentration) and changes in glucose, insulin, C-peptide, and glucagon during a mixed meal test.

ELIGIBILITY:
Inclusion Criteria:

* Males (Part 1 only) aged 18 to 55 years, and males and females (Part 2 only) aged 18 to 65 years inclusive at the time of signing informed consent
* Must agree to adhere to the contraception requirements
* Lean to overweight or obese but otherwise healthy males (Part 1 and 2) or nonpregnant, non-lactating females (Part 2 only)
* BMI of 22.0 to 32.0 kg/m2 for Part 1 and Part 2A, and a BMI of 27.0 to 35.0 kg/m2 for Part 2B and Part 2C, as measured at screening. Overweight or obese as assessed by BMI should be due to excess adipose tissue, as judged by the investigator
* Weight for males ≥70 kg (all parts), and for females ≥60 kg (Part 2 only) at screening

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Known or suspected hypersensitivity or allergy to paracetamol
* Presence or history of clinically significant cardiovascular, renal, hepatic, dermatological, respiratory, neurological, psychiatric, malignant, metabolic, endocrinological, haematological or venereal disorder, as judged by the investigator
* Presence or history of any clinically relevant gastrointestinal diseases or symptoms of gastrointestinal disorders potentially affecting interpretation of study data.
* Presence or history of diseases associated with impaired calcium homeostasis and/or increased bone turnover (e.g. Paget´s disease, osteoporosis)
* History of major depressive disorder within 2 years prior to screening
* Subjects unable to take paracetamol for any reason
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Subjects with tattoos or scars on the abdomen which may interfere with injection site assessments as determined by the investigator or delegate at screening
* Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed.
* HbA1c ≥48 mmol/mol (≥6.5%) and/or fasting plasma glucose ≥7.0 mmol/L at screening
* Part 2B only: Subjects with haemoglobin <LLN at screening and/or admission
* Prolongation of the QTcF over 450 msec for males and 470 msec for females or any other clinically significant abnormal ECG results as judged by the investigator
* Supine blood pressure (after ≥5 min rest) <90 mmHg or >150 mmHg (systolic) and/or <50 mmHg or >90 mmHg (diastolic)
* Heart rate (ECG-recorded after ≥5 min rest) <45 or >90 beats per minute
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
* Evidence of renal impairment at screening, as indicated by an estimated glomerular filtration rate (eGFR) of <70 mL/min/1.73m2
* Part 2 only: Females who are pregnant or lactating (all female subjects must have a negative highly sensitive urine or serum pregnancy test)
* Subjects who have received any investigational medicinal product (IMP) in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
* Subjects who have previously been administered IMP in this study
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies/vitamins in the 14 days before IMP administration.
* Paracetamol (up to 4 g per day) will be permitted except in the 48 h prior to the mixed meal tests on Day -1 and Day 4 (Part 1 Cohorts 2 to 6), Day 39 (Part 2A) and Day 81 (Part 2B) where paracetamol is not permitted.
* NSAIDs can be given at the discretion of the investigator to treat any AEs if necessary;
* Subject reports prior receipt of an amylin and/or calcitonin receptor agonist within the last 6 months
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week and in females >14 units per week
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Confirmed positive drugs of abuse test result at screening or admission
* Anticipated change in lifestyle (such as eating, exercise or sleeping pattern) during the trial and/or clinically significant body weight change (≥5% self-reported change) or comprehensive dieting attempts (e.g. participation in a weight reduction program or treatment with any medication indicated for weight management) within the last 90 days prior to screening
* Subjects who do not agree to consume the liquid mixed meal
* Male subjects with pregnant or lactating partners
* Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, that the investigator evaluates might jeopardise the subject's safety or compliance with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events (AE) incidence | from baseline (day 0) to end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  To provide safety information for GUB014295 by assessing: incidence of AEs categorized in System Organ Class (SOC) according to MedDRA (and evaluating severity and duration for SOC). No formal hypothesis will be tested in the study. Descriptive summaries for all safety safety data for all placebo, each active treatment and all active will be provided (including changes from baseline)
Safety - changes in vital signs | from baseline (day 0) to end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  To provide safety information for GUB014295 by assessing: Any changes from baseline for vital signs including: Blood pressure, Pulse/heart rate, oral temperature and respiratory frequency summarized as a ratio (baseline/end of trial).
  No formal hypothesis will be tested in the study. Descriptive summaries (as a relative change (ratio: 0 - 1) from day 0 to end of trial) for all safety safety data for all placebo, each active treatment and all active will be provided.
Safety - Safety laboratory parameters | From baseline (day 0) to end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  To provide safety information for GUB014295 by assessing a wide range of laboratory parameters within hematology, coagulation, clinical chemistry, virology, urinalysis.
  No formal hypothesis will be tested in the study. Descriptive summaries (as a relative change (ratio: 0 - 1) from day 0 to day end of trial)) for all safety safety data for all placebo, each active treatment and all active will be provided.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) - Tmax and Cmax | from dosing (day 0) until maximum concentration after final dose
  PK parameters: Tmax, (time of observed maximum concentration), Cmax (maximum observed concentration), for GUB014295.
Pharmacokinetic (PK) - area under the concentration curve (AUC) | From dosing (day 0) until end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  PK parameters:
  AUC(0-72) area under the curve for the GUB014295 measured from dosing, until 72 hours post dose, AUC(0-168) area under the curve for the GUB014295 measured from dosing, until 168 hours post dose, AUC(0-last) area under the curve for the GUB014295 measured from dosing, until the time of last measurable concentration, AUC(0-inf) area under the curve for the GUB014295 concentration from dosing, extrapolated until infinity.
Pharmacokinetic (PK) - T1/2 | from dosing (day 0) until end of trial (day 29)part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  PK parameters: T1/2: Terminal elimination half-life,
Pharmacokinetic (PK) - CL/F | from dosing (day 0) until end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  PK parameters:
  CL/F: Total body clearance (CL) calculated after single subcutaneous administration where F (fraction of bioavailability) is unknown,
Pharmacokinetic (PK) - Vz/F | From dosing (day 0) until end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  PK parameters:
  Vz/F: apparent volume of distribution (Vz) based on terminal phase calculated using AUC(0-inf) after a single subcutaneous administration where F (fraction of bioavailability) is unknown,

OTHER OUTCOMES:
Pharmacodynamic - body weight | From baseline (day 0) until end of trial (day 29) part 1, (day 64) part 2A, (day 120) part 2B and (day 127) in Part 2C
  Change in body weight (kg) from baseline to the end of the study. Descriptive summary for pharmacodynamic data (weight) including changes from baseline will be provided by all placebo and each active treatment.
Pharmacodynamic - liquid meal test incl. paracetamol (Part 1, Part 2A & Part 2B) | Before dosing (day -1) and day 4 part 1, day-1 and day 39 part 2A and day-1 and day 81 part 2B
  To investigate change in plasma concentration of glucose, insulin, C-peptide, glucagon and paracetamol in a paired liquid mixed meal test before (day-1) and after dosing (day 4 part 1, day-1 and day 39 part 2A and day-1 and day 81 part 2B) of a single dose of GUB014295. Descriptive summary (as a relative change (ratio: 0 - 1) from day -1 to day 4 part 1, day-1 and day 39 part 2A and day-1 and day 81 part 2B) for all pharmacodynamic data (glucose, insulin, C-peptide, glucagon and paracetamol) will be provided by all placebo and each active treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom